CLINICAL TRIAL: NCT06220721
Title: Reducing the Risk of Chronic Hypertension and Improving Vascular Function Following Preeclampsia
Acronym: REPAIR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Anna Palatnik, MD, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO00049909; 1R01HD112930-01A1 (NIH)
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Hypertension, Pregnancy-Induced
MeSH Terms: conditions — Hypertension, Pregnancy-Induced | interventions — Nifedipine

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- REPAIR ARM (Experimental): Intensive postpartum blood pressure control with nifedipine ER initiation at systolic blood pressure (SBP) ≥140 mmHg or diastolic blood pressure (DBP) ≥90 mmHg and maintaining blood pressure <140/90 mmHg during the first 6 weeks postpartum.
  Interventions: Drug: Nifedipine ER
- CONTROL ARM (Active Comparator): Usual care with nifedipine ER initiation at SBP ≥150 mmHg or DBP ≥100 mmHg and maintaining blood pressure <150/100 mmHg during the first 6 weeks postpartum.
  Interventions: Drug: Nifedipine ER

INTERVENTIONS:
Drug: Nifedipine ER — Initiation of nifedipine ER postpartum at randomly assigned threshold during the first 6 weeks postpartum.
  Other Names: Procardia XL; Adalat XL

SUMMARY:
The long-term goal of our work is to evaluate the effect of intensive postpartum blood pressure control on maternal cardiovascular health, risk of chronic hypertension, and reversal of vascular dysfunction generated by hypertensive disorders of pregnancy, thus attenuating the lifelong trajectory of cardiovascular disease risk.

DETAILED DESCRIPTION:
The REPAIR trial is a multicenter randomized controlled trial of 618 postpartum patients with hypertensive disorders of pregnancy randomized to intensive blood pressure control versus usual care during the first 6 weeks postpartum. The intervention group will receive intensive blood pressure (BP) control with nifedipine extended-release initiation when BP is ≥ 140/90 mmHg. The active control group will receive usual care with nifedipine ER initiation when BP is ≥ 150/100. The study will take place at two clinical sites: Medical College of Wisconsin (MCW) and Northwestern University (NU). All participants will undergo BP monitoring, cardiovascular function assessment, and collection of cardiovascular biomarkers at baseline, 6 weeks, and 12 months postpartum. Specifically, cardiac function and structure will be assessed with transthoracic echocardiogram, endothelial dysfunction with brachial artery flow-mediated dilation, and arterial stiffness with carotid-femoral pulse wave velocity. The primary outcome is the incident diagnosis of stage I hypertension at one year postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive disorders of pregnancy (HDP) diagnosis, specifically gestational hypertension, preeclampsia, eclampsia, or HELLP syndrome, according to ACOG guidelines
* Postpartum day 0-4
* Age ≥ 18 years
* Able to communicate in English or in Spanish
* Has an established OBGYN at an MCW or NU health system practice that has access to Epic electronic medical records.

Exclusion Criteria:

* Pre-gestational hypertension
* Type 1 or type 2 diabetes mellitus
* Admitted to intensive care unit at the time of screening
* Diagnosed with HDP during postpartum readmission after discharge from delivery hospitalization
* Getting discharged on the day of screening
* Known allergy or contraindication to nifedipine ER
* Inability or unwillingness to provide informed consent
* Already taking long-acting antihypertensive medication for standard care
* Maternal conditions that impact study outcomes: sickle cell disease, systemic lupus erythematosus

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 618 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Chronic hypertension | One year postpartum
  Diagnosis of chronic hypertension, defined as stage I hypertension with BP >130/80 mmHg

SECONDARY OUTCOMES:
Endothelial dysfunction | One year postpartum
  Brachial artery flow-mediated dilation will assess endothelial dysfunction.
Arterial stiffness | One year postpartum
  Carotid-femoral pulse wave velocity will assess arterial stiffness.
Cardiac structure and function | One year postpartum
  Transthoracic echocardiogram will assess cardiac structure and function.
Unplanned healthcare utilization | After birth through one year postpartum
  Unplanned hospital readmissions, emergency department visits, and clinic visits.
Composite severe maternal morbidity | After birth through one year postpartum
  Maternal core outcomes of preeclampsia using PMID: 32674052 reference.
Life's Essential 8 cardiovascular health score | After birth through one year postpartum
  The score (0-100) will be calculated using American Heart Association application.
Severe postpartum hypertension | After birth through one year postpartum
  Blood pressure >160/110 mmHg
ASCVD score | One year postpartum
  Lifetime risk calculated for subjects >20 years and 10-year risk calculated for subjects > 40 years.

OTHER OUTCOMES:
Serum biomarkers of cardiovascular risk | One year postpartum
  Soluble fms-like tyrosine kinase (sFlt-1), Lipoprotein (a), TNF-alpha, IL-6, NT-proBNP, CRP, high-sensitivity troponin
Breastfeeding initiation and duration | After birth through one year postpartum
  Assessed with Infant Feeding Practices Postnatal Questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Anna Palatnik, MD, Principal Investigator — Medical College of Wisconsin
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
After study closure, data will be deidentified, archived, and transmitted to the NICHD Data Specimen and Hub (DASH). Permission to transmit and store the data in DASH is included in the informed consent document.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Anticipated 6/30/2030
Access Criteria: The NICHD DASH Data Access Committee reviews all requests to access DASH data and biospecimens from identity-verified requesters to determine whether the proposed use is scientifically and ethically appropriate and does not conflict with constraints or research data use limitations identified by the institutions that submitted the research data or biospecimens.
URL: https://dash.nichd.nih.gov/resource/submission

REFERENCES:
- [Background] Duffy JMN, Cairns AE, Magee LA, von Dadelszen P, van 't Hooft J, Gale C, Brown M, Chappell LC, Grobman WA, Fitzpatrick R, Karumanchi SA, Lucas DN, Mol B, Stark M, Thangaratinam S, Wilson MJ, Williamson PR, Ziebland S, McManus RJ; International Collaboration to Harmonise Outcomes for Pre-eclampsia (iHOPE). Standardising definitions for the pre-eclampsia core outcome set: A consensus development study. Pregnancy Hypertens. 2020 Jul;21:208-217. doi: 10.1016/j.preghy.2020.06.005. Epub 2020 Jun 20. PMID 32674052
- [Background] Too G, Wen T, Boehme AK, Miller EC, Leffert LR, Attenello FJ, Mack WJ, D'Alton ME, Friedman AM. Timing and Risk Factors of Postpartum Stroke. Obstet Gynecol. 2018 Jan;131(1):70-78. doi: 10.1097/AOG.0000000000002372. PMID 29215510
- [Background] Wu P, Haththotuwa R, Kwok CS, Babu A, Kotronias RA, Rushton C, Zaman A, Fryer AA, Kadam U, Chew-Graham CA, Mamas MA. Preeclampsia and Future Cardiovascular Health: A Systematic Review and Meta-Analysis. Circ Cardiovasc Qual Outcomes. 2017 Feb;10(2):e003497. doi: 10.1161/CIRCOUTCOMES.116.003497. Epub 2017 Feb 22. PMID 28228456
- [Background] Parikh NI, Gonzalez JM, Anderson CAM, Judd SE, Rexrode KM, Hlatky MA, Gunderson EP, Stuart JJ, Vaidya D; American Heart Association Council on Epidemiology and Prevention; Council on Arteriosclerosis, Thrombosis and Vascular Biology; Council on Cardiovascular and Stroke Nursing; and the Stroke Council. Adverse Pregnancy Outcomes and Cardiovascular Disease Risk: Unique Opportunities for Cardiovascular Disease Prevention in Women: A Scientific Statement From the American Heart Association. Circulation. 2021 May 4;143(18):e902-e916. doi: 10.1161/CIR.0000000000000961. Epub 2021 Mar 29. PMID 33779213
- [Background] Hauspurg A, Lemon L, Cabrera C, Javaid A, Binstock A, Quinn B, Larkin J, Watson AR, Beigi RH, Simhan H. Racial Differences in Postpartum Blood Pressure Trajectories Among Women After a Hypertensive Disorder of Pregnancy. JAMA Netw Open. 2020 Dec 1;3(12):e2030815. doi: 10.1001/jamanetworkopen.2020.30815. PMID 33351087
- [Background] Shahul S, Tung A, Minhaj M, Nizamuddin J, Wenger J, Mahmood E, Mueller A, Shaefi S, Scavone B, Kociol RD, Talmor D, Rana S. Racial Disparities in Comorbidities, Complications, and Maternal and Fetal Outcomes in Women With Preeclampsia/eclampsia. Hypertens Pregnancy. 2015 Nov;34(4):506-515. doi: 10.3109/10641955.2015.1090581. Epub 2015 Dec 4. PMID 26636247
- [Background] Levine L, Arany Z, Kern-Goldberger A, Koelper N, Lewey J, Sammel MD, Elovitz MA, Ky B. Soluble Flt1 levels are associated with cardiac dysfunction in Black women with and without severe preeclampsia. Hypertens Pregnancy. 2021 Feb;40(1):44-49. doi: 10.1080/10641955.2020.1861462. Epub 2020 Dec 20. PMID 33345653
- [Background] Grand'Maison S, Pilote L, Okano M, Landry T, Dayan N. Markers of Vascular Dysfunction After Hypertensive Disorders of Pregnancy: A Systematic Review and Meta-Analysis. Hypertension. 2016 Dec;68(6):1447-1458. doi: 10.1161/HYPERTENSIONAHA.116.07907. Epub 2016 Oct 17. PMID 27754864
- [Background] Lane-Cordova AD, Khan SS, Grobman WA, Greenland P, Shah SJ. Long-Term Cardiovascular Risks Associated With Adverse Pregnancy Outcomes: JACC Review Topic of the Week. J Am Coll Cardiol. 2019 Apr 30;73(16):2106-2116. doi: 10.1016/j.jacc.2018.12.092. PMID 31023435
- [Background] Weissgerber TL, Milic NM, Milin-Lazovic JS, Garovic VD. Impaired Flow-Mediated Dilation Before, During, and After Preeclampsia: A Systematic Review and Meta-Analysis. Hypertension. 2016 Feb;67(2):415-23. doi: 10.1161/HYPERTENSIONAHA.115.06554. Epub 2015 Dec 28. PMID 26711737
- [Background] Hirshberg A, Downes K, Srinivas S. Comparing standard office-based follow-up with text-based remote monitoring in the management of postpartum hypertension: a randomised clinical trial. BMJ Qual Saf. 2018 Nov;27(11):871-877. doi: 10.1136/bmjqs-2018-007837. Epub 2018 Apr 27. PMID 29703800
- [Background] Lopes Perdigao J, Hirshberg A, Koelper N, Srinivas SK, Sammel MD, Levine LD. Postpartum blood pressure trends are impacted by race and BMI. Pregnancy Hypertens. 2020 Apr;20:14-18. doi: 10.1016/j.preghy.2020.02.006. Epub 2020 Feb 26. PMID 32143061
- [Background] Stuart JJ, Tanz LJ, Rimm EB, Spiegelman D, Missmer SA, Mukamal KJ, Rexrode KM, Rich-Edwards JW. Cardiovascular Risk Factors Mediate the Long-Term Maternal Risk Associated With Hypertensive Disorders of Pregnancy. J Am Coll Cardiol. 2022 May 17;79(19):1901-1913. doi: 10.1016/j.jacc.2022.03.335. PMID 35550687
- [Background] Whelton PK, Carey RM, Aronow WS, Casey DE Jr, Collins KJ, Dennison Himmelfarb C, DePalma SM, Gidding S, Jamerson KA, Jones DW, MacLaughlin EJ, Muntner P, Ovbiagele B, Smith SC Jr, Spencer CC, Stafford RS, Taler SJ, Thomas RJ, Williams KA Sr, Williamson JD, Wright JT Jr. 2017 ACC/AHA/AAPA/ABC/ACPM/AGS/APhA/ASH/ASPC/NMA/PCNA Guideline for the Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2018 May 15;71(19):e127-e248. doi: 10.1016/j.jacc.2017.11.006. Epub 2017 Nov 13. No abstract available. PMID 29146535
- [Background] Lloyd-Jones DM, Allen NB, Anderson CAM, Black T, Brewer LC, Foraker RE, Grandner MA, Lavretsky H, Perak AM, Sharma G, Rosamond W; American Heart Association. Life's Essential 8: Updating and Enhancing the American Heart Association's Construct of Cardiovascular Health: A Presidential Advisory From the American Heart Association. Circulation. 2022 Aug 2;146(5):e18-e43. doi: 10.1161/CIR.0000000000001078. Epub 2022 Jun 29. PMID 35766027